CLINICAL TRIAL: NCT05042011
Title: Role of mHealth-based Interventions Including Social Media to Improve Childhood Immunization Coverage During COVID 19 Pandemic in Pakistan: Qualitative Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Dr Abdul Momin Kazi, Assistant Professor, Aga Khan University
Other Study IDs: 2020-5316-14620
Record Dates: First submitted 2021-03-19; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: mHealth; Social Media; Vaccine Hesitancy; Covid19
Keywords: Covid19; childhood routine immunization (CRI); mHealth; social media
MeSH Terms: conditions — Vaccination Hesitancy; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to improve routine immunization uptake during COVID-19 pandemic, and to understand the perceptions and barriers related to vaccine hesitancy and coverage during COVID 19 and to explore the need for COVID-19 vaccination, separately and as a part of routine immunization, the investigators will be using qualitative methodology to explore and understand the role of mHealth and social media interventions, that are most suitable in Pakistani context to improve vaccination coverage during COVID-19 pandemic.

DETAILED DESCRIPTION:
The application of information and communication technologies (through such digital health methods as SMS, phone calls and automated calls, smartphone apps and wearable technology) has paved the way for modification of health-related knowledge and bring in the behavior change and practices to decrease vaccine hesitancy and improve immunization uptake. Mass and social media are influential in the dissemination of information regarding the COVID-19 pandemic, as well as the development and use of vaccines, not only for COVID-19 but also CRI. However, the same low-cost/free and accessible methods (social media platforms) that enable low/middle-income populations to communicate, connect and access information can also be the main factor in the distribution and prevalence of unregulated, unverified misinformation. In particular, the anti-vaccination movement, which has been identified as a major factor for vaccine hesitancy is the result of spreading misinformation through these same social media platforms.

In light of the current pandemic and distancing measures, CRI coverage is adversely affected as caregivers avoid tertiary care hospitals or primary health centers. This has further increased the risk of outbreak for vaccine-preventable diseases, as well as economic burden due to morbidity and mortality and delay in caregiver getting back to work. A recent survey by an international consortium also illustrated a decline in vaccination coverage across all milestone age groups, except for vaccines administered at birth in hospital like Hepatitis B. Hence due to reduced vaccination rates, various countries are experiencing outbreaks of previously controlled diseases globally like measles, rubella, tuberculosis, and rotavirus, and has even caused new mutated strains of polio to reemerge. However, for the first time in almost three decades there has been the significant decrease in the coverage of DPT3 vaccine dose.

Pakistan is identified as a LMIC with high vaccine hesitancy and is third among countries with the most unvaccinated/under-vaccinated children. It ranks fourth in global child mortality, with 60% of deaths due to infectious diseases that are vaccine-preventable. The EPI coverage for fully immunized children were estimated to be 65% and 88% at national level respectively in the past two survey reports. However, rates for Sindh province are even lower with fully immunized children rates of 39% and 80% respectively. Further Pakistan is among three polios endemic country and among top 5 countries with the most unvaccinated and under-vaccinated children. With further decrease in immunization rates due to current pandemic, vaccination coverage has only plummeted all time low coverage further due to disruption in vaccination services and demand, causing new outbreaks of previously controlled diseases like new polio strains, measles and rubella. Hence it is eminent to explore new strategies included mhealth and social media to bring in the behavior change in order to improve vaccine uptake. In addition, it is also important to understand the perceptions and barriers related to vaccine hesitancy and coverage during COVID 19 and come up with strategies to finalize our interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Caregivers of children less than one year of age will be enrolled from HDSS sites.
2. Health care providers including (doctors, nurses, pharmacists, LHVs, Vaccinators, LHWs, etc.) will also be recruited from these sites.

Exclusion Criteria:

1. The exclusion criteria include the children from outside the health demographic surveillance system (HDSS) area and if the family does not plan to stay in the catchment area.
2. Health care providers will be excluded who are from outside the HDSS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers of children less than one year of age and Health care providers working inthe HDSS sites.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Hesitancy towards childhood routine immunization (Interview) | 2 months
  Questions To understand the perceptions and barriers related to routine immunization during COVID-19 pandemic
COVID-19 vaccine hesitancy (Interview) | 2 months
  Questions To understand the perceptions and barriers related to COVID-19 vaccine for adults and as part of routine immunization
Role of mHealth and social media (Interview) | 2 months
  Questions To understand the role of mHealth and social media in improving childhood immunization coverage and COIVD-19 vaccine during COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan